CLINICAL TRIAL: NCT05551325
Title: Reestablishing Sleep and Circadian Alignment in Medically Critically Ill Patients Via a Mechanistic Randomized Controlled Trial (RCT) of an Intensive Care Unit (ICU) Sleep Chronobundle
Brief Title: Reestablishing Sleep and Circadian Alignment in Medical Intensive Care Unit (MICU) Patients Via a Mechanistic RCT of an Sleep Chronobundle
Acronym: ReAlign-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000033373; 1R01HL163659-01A1 (NIH)
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness; Sleep Deprivation; Circadian Rhythm Sleep Disorder, Unspecified
Keywords: critical illness; sleep deficiency; circadian misalignment
MeSH Terms: conditions — Critical Illness; Sleep Deprivation; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of patients to control or intervention
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention participants, care providers, and investigators will be able to ascertain group assignment.
  Primary and secondary outcome assessors of urine 6-sulfatoxymelatonin levels, sleep scoring, and glucose levels via continuous glucose monitoring will be masked from group assignment.
  Exploratory outcome assessors will be able to ascertain group assignment as they will be at the patient's bedside or in the medical record during the process of recording outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual ICU care.
- Chronobundle (Experimental): The chronobundle will include bright daytime light, time-restricted intermittent feeding, enhanced exercise/mobility, and overnight sleep promotion.
  Interventions: Other: Chronobundle - light; Other: chronobundle - feeding; Other: chronobundle - mobility; Other: chronobundle - sleep

INTERVENTIONS:
Other: Chronobundle - light — Bright daytime light from 09:00 to 13:00 starting on day 1. The light will be 10,000 lux at 12" and provide a minimal intensity of 1,250 lux at the angle of the eye (30" to 36" distance). The light has a temperature of 5,000 Kelvin indicating a high blue wavelength content which should maximize circadian effects (validated device Sunbox Lighting, Maryland). Following the 09:00 to 13:00 bright light, the room lights will remain on and the curtains will remain open to maximize daytime light exposure while not decreasing bright light tolerance.
  Arms: Chronobundle
Other: chronobundle - feeding — For patients receiving enteral feeds, time-restricted (daytime) intermittent feeding will include 4 meals delivered at 08:00, 12:00, 16:00 and 20:00. Each meal will include one-fourth of the recommended daily tube feed volume.
  Arms: Chronobundle
Other: chronobundle - mobility — While in the MICU, exercise/mobility sessions led by physical therapy or occupational therapy providers will occur twice daily between 09:00 and 16:00 (i.e., one additional session beyond usual care); intensity will be determined by clinical status and documented in the chart by our physical therapy service. Patients in other hospital locations (e.g., general medical ward post-MICU discharge) will receive one additional session beyond usual care via a study staff-led exercise/mobility session; intensity will be determined by clinical status.
  Arms: Chronobundle
Other: chronobundle - sleep — Overnight sleep promotion will occur between 22:00 and 06:00 with a more restricted sleep period between 00:00 and 04:00. This will be achieved by rescheduling non-urgent care. There will be no changes to urgent care. Additionally, room lights will be dimmed, curtains drawn, and room doors closed. Television screens will be fitted with blue light-blocking filters.
  Arms: Chronobundle

SUMMARY:
More than 5 million patients are admitted to the intensive care unit every year in the United States; most of these patients experience profound sleep and circadian disruption. Promotion of circadian alignment (i.e., alignment of the body's clocks) would make it possible to strategically schedule behaviors such as sleep and eating at normal body clock times, which is predicted to improve sleep quality and metabolic function. This project will test the ability of a sleep chronobundle (i.e., sleep promotion and circadian treatment bundle) to normalize circadian alignment and subsequently test if this realignment also improves sleep and metabolism.

DETAILED DESCRIPTION:
An evidence-based treatment that simultaneously addresses intensive care unit (ICU) sleep and circadian disruption (SCD) is desperately needed. Such treatment is needed because patients admitted to the ICU are at high risk for adverse outcomes resulting directly from acute SCD. It is well established among healthy controls that acute SCD is associated with immediate negative consequences such as metabolic, cognitive, cardiovascular, respiratory, skeletal muscle, and immune dysfunction. Normalization of sleep and circadian processes improves these dysfunctions. In the ICU, sleep and circadian processes cannot be segregated, and there are likely several overlapping domains of SCD (e.g., sleep duration, timing, architecture, and continuity, and circadian alignment and amplitude). Thus, a bundled approach to sleep and circadian promotion holds the most promise for reversing SCD, normalizing broader physiologic disruptions, and improving ICU outcomes.

To date, ICU sleep promotion bundles have had limited success in documenting improved sleep, and sleep bundles have commonly ignored circadian disruption and circadian-based sleep promotion strategies. This is a critical gap. Translation of circadian principles to ICU sleep promotion is essential because alignment between biologic and clock time allows for subsequent strategic scheduling of behaviors, for example, scheduling sleep promotion during the biologic night to improve sleep duration and quality. In addition, circadian alignment has broader physiologic implications and related potential to improve function across a wide variety of organ systems, for example, scheduling eating during the biologic day to improve glucose tolerance. Investigations to date have not tested the effect of a multifaceted intervention that includes promotion of both circadian alignment via photic and nonphotic zeitgebers and overnight sleep via non-pharmacologic strategies (sleep chronobundle).

The overall objective of this project is to test whether a sleep chronobundle, including daytime bright light, time-restricted daytime feeding, increased daytime mobility, and overnight sleep promotion mitigates ICU SCD. A mechanistic randomized controlled trial will be used to test our central hypotheses that a sleep chronobundle will (1) align biologic and clock day-night; (2) overlap behaviors (e.g., sleeping and eating) correctly with biologic time periods; and therefore (3) improve sleep and metabolic processes in the ICU. The focus of this study is on sleep and glucose metabolism metrics because of their high relevance to critical illness.

ELIGIBILITY:
Inclusion:

* Critically ill patients admitted to the MICU who require mechanical ventilation, noninvasive ventilation, high flow nasal cannula, or vasopressor support and who remain on qualifying support as of 09:00 on study randomization day. Randomization will occur on the second or third calendar day following MICU admission. MICU admission must have occurred within 24 hours of hospital admission.
* Age greater than or equal to 18 years old.

Exclusion:

* Not expected to remain in the MICU for at least 48 hours post-randomization.
* Imminently dying or with a hospice status.
* At significant risk for pre-existing circadian abnormalities including: (1) severe chronic brain injury (injury greater than 30 days ago resulting in the inability to live independently); (2) acute brain injury of any severity that is reasonably expected to impact the central circadian clock (e.g., cardiac arrest); (3) documented circadian disorder (<1% population) or blind/disease of the optic nerve; (4) current or recent (last 1 year) shiftwork; and (5) homelessness, incarceration, or institutionalization.
* At elevated risk of aspiration due to structural or functional abnormality of the gastrointestinal tract OR fed via enteral nutrition (e.g., "tube feeds") prior to ICU admission.
* Admitted to the ICU for treatment of diabetic ketoacidosis or hyperosmolar state; this diagnosis will be established via review of the medical record for a description of diabetes in the past medical history or the presence of diabetes medication on the confirmed home medication list AND hyperglycemia attributed to diabetic ketoacidosis or diabetic hyperosmolar state by the admitting care team in their written assessment of the patient.
* Having a history of hypoglycemia without documented full neurological recovery; this diagnosis will be established via review of the patient's past medical history in the medical record;
* Having a history suggesting an abnormally high risk of suffering hypoglycemia (e.g., known insulin secreting tumor, history of unexplained or recurrent hypoglycemia or fulminant hepatic failure); this diagnosis will be established via review of the patient's past medical history in the medical record.
* Admitted due to complications of a suicide attempt.
* Admitted due to an acute drug overdose or active alcohol withdrawal.
* Positive for SARS-CoV.

Urine 6-sulfatoxymelatonin measures will be considered for all patients who make sufficient urine and have an appropriate bladder catheter in place during the indicated time points. However, we will exclude patients from urine measures if they have a history or positive test for any known disease or illness that would categorize biological samples as BSL3 or higher. This includes HIV, West Nile virus, Monkeypox, and Mycobacterium tuberculosis (TB).

Note: Patients who leave the MICU within 24 hours of randomization are excluded from further study activities. Patients who leave the MICU between 24 and 48 hours post-randomization continue all study activities but will not be included in the primary analysis. Patients who remain in the MICU for at least 48 hours post-randomization will continue all study activities and be included in the primary analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2028-06-29 (Estimated); Study Completion 2028-06-29 (Estimated)

PRIMARY OUTCOMES:
Circadian alignment based on diurnal heart rate variation | post-treatment, 72 hours
  Individual heart rate nadir compared to population normal nadir of 04:00. Maximum difference +/- 12 hours.

SECONDARY OUTCOMES:
Urine 6-sulfatoxymelatonin acrophase change from normal | post-treatment, 72 hours
  Individual urine 6-sulfatoxymelatonin acrophase compared to population normal acrophase of 03:30. Maximum difference +/- 12 hours. Urine 6-sulfatoxymelatonin measures will be completed for all patients who make sufficient urine and have an appropriate bladder catheter in place during the indicated time points.
Urine 6-sulfatoxymelatonin acrophase absolute time | post-treatment, 72 hours
  Clock time of individual urine 6-sulfatoxymelatonin acrophase. Urine 6-sulfatoxymelatonin measures will be completed for all patients who make sufficient urine and have an appropriate bladder catheter in place during the indicated time points.
Urine 6-sulfatoxymelatonin acrophase change from day 1 to day 4 | Day 1 and post-treatment, 72 hours
  Change in individual urine 6-sulfatoxymelatonin acrophase between day 1 observation and day 4 observation period (after 72 hours intervention). Urine 6-sulfatoxymelatonin measures will be completed for all patients who make sufficient urine and have an appropriate bladder catheter in place during the indicated time points.
Overnight sleep duration | post-treatment, 72 hours
  Minutes of sleep from 22:00 to 05:59 as measured by NoxA1 portable polysomnography (PSG) device.
Overnight Rapid Eye Movement (REM) proportion | post-treatment, 72 hours
  Proportion of Stage REM sleep from 22:00 to 05:59 as measured by NoxA1 portable polysomnography device.
Overnight non-rapid eye movement stage 3 (NREM3) proportion | post-treatment, 72 hours
  Proportion of Stage NREM3 sleep from 22:00 to 05:59 as measured by NoxA1 portable polysomnography device.
Overnight arousal index (continuity) | post-treatment, 72 hours
  Number of arousals per hour of sleep from 22:00 to 05:59 as measured by NoxA1 portable polysomnography device.
Daytime sleep duration | post-treatment, 72 hours
  Minutes of sleep from 06:00 to 21:59 as measured by NoxA1 portable polysomnography device.
Daytime REM proportion | post-treatment, 72 hours
  Proportion of Stage REM sleep from 06:00 to 21:59 as measured by NoxA1 portable polysomnography device.
Daytime NREM3 proportion | post-treatment, 72 hours
  Proportion of Stage NREM3 sleep from 06:00 to 21:59 as measured by NoxA1 portable polysomnography device.
Daytime arousal index (continuity) | post-treatment, 72 hours
  Number of arousals per hour of sleep from 06:00 to 21:59 as measured by NoxA1 portable polysomnography device.
Biologic night sleep duration | post-treatment, 72 hours
  Minutes of sleep during biologic night (melatonin onset to offset) as measured by NoxA1 portable polysomnography device. Biologic night determination will be completed for all patients who make sufficient urine and have an appropriate bladder catheter in place during the indicated time points.
Biologic night REM proportion | post-treatment, 72 hours
  Proportion of Stage REM sleep during biologic night (melatonin onset to offset) as measured by NoxA1 portable polysomnography device. Biologic night determination will be completed for all patients who make sufficient urine and have an appropriate bladder catheter in place during the indicated time points.
Biologic night NREM3 proportion | post-treatment, 72 hours
  Proportion of Stage NREM3 sleep during biologic night (melatonin onset to offset) as measured by NoxA1 portable polysomnography device. Biologic night determination will be completed for all patients who make sufficient urine and have an appropriate bladder catheter in place during the indicated time points.
Biologic night arousal index (continuity) | post-treatment, 72 hours
  Number of arousals per hour of sleep during biologic night (melatonin onset to offset) as measured by NoxA1 portable polysomnography device. Biologic night determination will be completed for all patients who make sufficient urine and have an appropriate bladder catheter in place during the indicated time points.
Atypical sleep | post-treatment, 72 hours
  Presence of atypical sleep on polysomnography recording, characterized by δ waves without cyclic organization, the absence of K-complexes and sleep spindles, and unusual sleep stage transitions.
Glucose tolerance | post-treatment, 72 hours
  Area under the curve per 24 hour period of continuous glucose monitoring.

OTHER OUTCOMES:
Exploratory - Days without Delirium or Coma | post-treatment, 14 days post randomization
  Days alive and without delirium or coma out of the 14 days post randomization
Exploratory - Ventilator Free Days | post-treatment, 28 days post randomization
  Days alive and ventilator free out of 28 days post-randomization.
Exploratory - Time to ICU Discharge | post-treatment
  Days to ICU discharge post-randomization.
Exploratory - Time to Hospital Discharge | post-treatment
  Days to hospital discharge post-randomization.
Exploratory - Mortality | post-treatment, 30 days post-randomization
  Mortality at 30 days post-randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa P Knauert, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital Medical Intensive Care Unit (YNHH MICU) at St Raphael's Campus, New Haven, Connecticut
  - Yale New Haven Hospital Medical Intensive Care Unit (YNHH MICU) at York Street, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No